CLINICAL TRIAL: NCT06186414
Title: An Open-Label, Multicenter Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SIM0237 Alone or in Combination with BCG in Non-Muscle-Invasive Bladder Cancer
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SIM0237 Alone or in Combination with BCG in NMIBC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: Shanghai Xianxiang Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SIM0237-102
Record Dates: First submitted 2023-12-07; First posted 2024-01-02 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-06

CONDITIONS: Non-Muscle-Invasive Bladder Cancer (NMIBC)
Keywords: NMIBC
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Dose escalation-mono (Experimental): BCG-unresponsive high-risk NMIBC, receiving SIM0237 monotherapy intravesically.
  Interventions: Drug: SIM0237
- Dose escalation-combo (Experimental): BCG-unresponsive high-risk NMIBC, receiving SIM0237 and BCG intravesically.
  Interventions: Drug: SIM0237 and BCG
- Dose expansion-Cohort 1 (Experimental): BCG-unresponsive CIS, receiving SIM0237 monotherapy intravesically.
  Interventions: Drug: SIM0237
- Dose expansion-Cohort 3 (Experimental): BCG-unresponsive CIS, receiving SIM0237 and BCG intravesically.
  Interventions: Drug: SIM0237 and BCG
- Dose expansion-Cohort 4 (Experimental): BCG-unresponsive high-risk Ta or T1, receiving SIM0237 and BCG intravesically.
  Interventions: Drug: SIM0237 and BCG
- Dose expansion-Cohort 2 (Experimental): BCG-unresponsive high-risk Ta or T1, receiving SIM0237 monotherapy intravesically.
  Interventions: Drug: SIM0237

INTERVENTIONS:
Drug: SIM0237 — Several dose levels of SIM0237 will be administered as a single agent for evaluation
  Arms: Dose escalation-mono
Drug: SIM0237 and BCG — Several dose levels of SIM0237 will be administered in combination with a fixed dose of BCG for evaluation
  Arms: Dose escalation-combo
Drug: SIM0237 — RD level of SIM0237 will be administered as a single agent for evaluation
  Arms: Dose expansion-Cohort 1; Dose expansion-Cohort 2
Drug: SIM0237 and BCG — RD level of SIM0237 will be administered in combination with a fixed dose of BCG for evaluation
  Arms: Dose expansion-Cohort 3; Dose expansion-Cohort 4

SUMMARY:
This is an open-label, multicenter phase 1 study to evaluate the safety, efficacy, and pharmacokinetics (PK) characteristics of SIM0237 alone or in combination with bacillus Calmette-Guerin (BCG) in participants with Non-Muscle-Invasive Bladder Cancer (NMIBC)

DETAILED DESCRIPTION:
The study starts with a dose escalation part followed by a dose expansion part. The primary objective of the dose escalation part is to evaluate the safety and tolerability of SIM0237 alone or in combination with BCG, and determine the recommended dose(s) (RD). The primary objective of the dose expansion part is to evaluate the preliminary efficacy of SIM0237 alone or in combination with BCG.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* ≥ 18 years of age, male or female.
* • Histologically confirmed presence of BCG-unresponsive CIS (with or without Ta or T1 disease) or histologically confirmed presence of BCG-unresponsive high-grade Ta or T1 disease. Histologic confirmation of urothelial carcinoma (mixed histology tumors allowed if urothelial histology is predominant histology).
* Dose escalation phase: BCG-unresponsive high-risk NMIBC.
* Dose expansion phase: a) Cohorts 1 and 3: BCG-unresponsive CIS (with or without Ta or T1 disease); b) Cohort 2 and 4: BCG-unresponsive high-risk Ta or T1 disease.
* Absence of resectable disease after transurethral resection (TURBT) procedures [residual carcinoma in situ (CIS) acceptable]. patients with T1 tumors must undergo repeat resection and pathological test if initial pathological test sample did not include muscularis propria, to ensure the inclusive of muscularis propria and the absence of invasive tumor.
* Not suitable for or unwilling to undergo radical cystectomy.
* ECOG performance status of 0, 1or 2.
* Life expectancy ≥ 2 years.
* Adequate hematologic and organ function.
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test. WOCBP and male subjects agree to use adequate contraception.
* Tumor tissue (archival or fresh) for biomarker analysis.

Exclusion Criteria:

* • Subjects received TURBT or other surgical treatment for bladder lesions or pelvic radiotherapy or interventional therapy within 2 weeks prior to the first dose.
* Previous treatment with: a) IL-15 or IL-2; b) immune checkpoint inhibitors (such as anti-PD-1 or PD-L1 antibodies), ADCs, chemotherapies, oncolytic viruses, BCG or other anti-tumor treatments, unless there is clear evidence of disease persistence/recurrence/progression after the above treatments and beyond 4 weeks prior to the first dose; c) Chinese herbal medicine treatment beyond 2 weeks prior to the first dose is allowed; d) A single immediate instillation of chemotherapy within 4 weeks prior to the first dose is allowed; e) intravesical instillation of mucosal protective agents (e.g., sodium hyaluronate) are allowed.
* Subject is participating in an investigational drug or investigational device study.
* Subjects have not recovered from AEs caused by previous anti-tumor treatment.
* History/evidence of prior muscle-invasive, locally advanced, metastatic bladder cancer or upper urinary tract (kidney, renal pelvis, ureter) and prostatic urethral tumors; or evidence of Ta/T1/CIS urothelial transitional cell carcinoma outside the bladder (urethra, ureter, renal pelvis) during the screening period.
* Patients with other malignancies within 5 years before the first dose.
* Any active infection or urinary tract infection requiring systemic treatment by intravenous infusion within 2 weeks before the first dose.
* Subjects with clinically significant cardiovascular disease within 6 months before the first dose of study treatment.
* Known human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS).
* Active or chronic hepatitis B or hepatitis C infection.
* Known or suspected active autoimmune diseases.
* Concurrent use of any other anticancer therapy or chronic use of systemic corticosteroids at immunosuppressive doses (more than 10 mg/day prednisone or equivalent).
* History of pneumonitis or interstitial lung disease or severe obstructive pulmonary disease that requires oral or intravenous steroids to help recover.
* Known to be allergic or intolerant to study drugs, monoclonal antibodies, excipients; or allergic or intolerant to BCG (only for subjects receiving combined BCG therapy)
* Subjects discontinued prior BCG treatment due to AEs such as toxemia, systemic infection, or urinary incontinence (only for subjects receiving combined BCG therapy).
* History of allogeneic organ transplantation or graft-versus-host disease.
* Any live vaccines within 4 weeks before the first dose.
* Known mental illness or substance abuse that would interfere with trial complies.
* Subject is pregnant or lactating, or is expected to become pregnant or parent a child during the planned study period.
* Other conditions that investigators consider inappropriate for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Dose escalation:Dose limited toxicity (DLT) | DLT observation period (up to 21 days)
Dose escalation: Percentage of participants experiencing treatment-emergent adverse events (TEAEs) | through study completion, an average of 5 years
  Incidence and severity of adverse events (AEs) and serious adverse events(SAEs),and lab abnormalities
Dose expansion:Complete response (CR) rate at Month 3 | through study completion, an average of 5 years
  Complete response (CR) rate at of Cohort 1 and Cohort 3
Dose escalation: Percentage of participants experiencing AE related dose interruptions and dose delays, dose intensity | through study completion, an average of 5 years
  Occurrence of AE related dose interruptions, dose delays and dose intensity

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Haerbin, Heilongjiang
  - Henan Cancer Hospital Affiliated Cancer Hospital of Zhengzhou University, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medcial University, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No